CLINICAL TRIAL: NCT00278759
Title: Unclogging the Pediatric Emergency Room: Impact of Rapid Viral Diagnostics. A Randomized Controlled Trial of Decision Making Based Upon Early (at Triage) Rapid Diagnosis of Respiratory Viral Infections (VIRAP) in Children 3-36 Months of Age Presenting to the Emergency Department (ED) With a Flu-Like Illness.
Brief Title: Unclogging the Pediatric Emergency Room: Impact of Rapid Viral Diagnostics
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Collaborators: Michael Smith Foundation for Health Research (Other)
Responsible Party: Dr. Eva Thomas, University of British Columbia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: C05-0501
Record Dates: First submitted 2006-01-16; First posted 2006-01-18 (Estimated); Last update posted 2009-02-19 (Estimated); Status verified 2008-08

CONDITIONS: Respiratory Infection
Keywords: rapid viral diagnosis; respiratory infection; pediatric emergency department; febrile respiratory infection
MeSH Terms: conditions — Respiratory Tract Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Nasopharyngeal washing for viral antigen detection by immunofluorescence initiated early in ED visit. — See Detailed Description.

SUMMARY:
Acute respiratory tract infections are among the most common problems of childhood, particularly among infants and children younger than 3 years, and account for most antibiotic prescriptions to children. Most of these infections are self-limited and do not require medical intervention; however, the symptoms overlap significantly with those of severe viral or bacterial infections. At the hospital Emergency Department (ED), medical assessment, prescription of antibiotics (unnecessarily if the infection is viral), and a series of investigations (e.g., blood work, X-rays) often take place before a decision on patient management and possible hospital admission can be made. Such procedures lead to intense use of human health resources (nursing, laboratory and radiology staff) and hospital facilities.

The literature suggests that a prompt single viral diagnosis improves decision-making. To our knowledge, no-one has performed a controlled trial to examine the impact of a rapid, multi-viral detection test like VIRAP, or the impact of the timing of such a test, on management of children with flu-like illnesses in the ED.

Our objective is to determine if use of our new viral detection program, VIRAP, for rapid testing for viral respiratory infections right after triage will improve patient management and resource use in the ED. We will test the hypothesis that availability of VIRAP at triage to support rapid diagnosis of viral infection in children at BCCH will (i) reduce the waiting time in the ED; (ii) improve decision making regarding diagnostic investigations and specimen collection; and (iii) decrease antibiotic prescriptions.

Study completed and manuscript accepted for publication in the Journal of Pediatrics.

DETAILED DESCRIPTION:
Description of Project:

Background: Acute viral respiratory tract infections are among the most common infectious problems of childhood during the first five years of life, particularly among infants younger than 2 years of age. Although the majority of these infections does not require medical attention and are self-limited in nature, worried parents commonly bring their children to the emergency department (ED) for evaluation (average 2500 children/winter). EDs are choke points in the health care system, especially at the peaks of the annual influenza season and respiratory syncytial virus (RSV) season. Without a prompt specific viral diagnosis in a child presenting to the ED with a febrile respiratory illness, after being seen by a physician, a child may have to undergo a constellation of precautionary diagnostic tests (septic work up, CXR) and be prescribed antibiotics unnecessarily. These interventions lead to prolonged ED stays (average 180min +/-120 min), intense use of human health resources (nursing, laboratory and radiology staff) resulting in significant cost both direct and indirect to the health care system, as well as time lost to the children and their families and contribute to antimicrobial resistance. The precise etiology of these viral infection episodes can be determined through the use of rapid screening program such as VIRAP (nasopharyngeal washing for rapid direct viral antigen detection via immunofluorescence). At the moment VIRAP is a physician ordered test, done only after the child has been seen by the physician, usually after the child has already been waiting for a significant length of time, then has to wait further for the results of the test.

Hypothesis: Rapid diagnosis of viral infection through VIRAP initiated by a nurse at triage wit results available for ED physician time of assessment may influence decision making with respect to additional investigations therefore reduce the amount of waiting time in the ED, as well as decrease antibiotic prescriptions. This would ultimately result in improved effectiveness of service provision for children with febrile respiratory illnesses and in turn shorten waiting time for all children in the ED. Health care cost reduction by minimising unnecessary diagnostic tests being performed and antibiotic prescription are also expected.

Study design: We propose to conduct a single centre, open label, randomized controlled trial comparing outcomes of patients undergoing VIRAP at triage vs routine ED admission protocol. During the months of December 2005 to April, and again Dec2006 to April 2007, eligible patients based on our inclusion and exclusion will be enrolled at triage and randomized in a 1:1 ratio to either undergo NPW for VIRAP and have the result available to the treating physician at time of assessment or routine admitting protocol to the ED and await physician assessment without prior investigation.

Criteria: Patients age 3-36 months admitted to the BCCH ED with fever(≥38.5 0C measured in ED or documented by the accompanying parent) and at least one of: cough, runny nose, nasal congestion and sore throat will be eligible for enrolment. Excluded from the study will be patients who are immuno-compromised, who have underlying chronic severe respiratory conditions (cystic fibrosis, bronchopulmonary dysplasia) or chronic heart conditions (uncorrected cyanotic heart lesions, prosthetic valves), who have had prior assessment in our ED department for the current illness. Only one child per family can be enrolled.

End points: The duration of stay in ED (from assessment to discharge, including time waiting for investigations and review of results by the physician) is the primary endpoint. Secondary endpoints include whether any investigations following the assessment (blood test, radiographs or urine tests) were ordered and whether study patients were prescribed antibiotics.

ELIGIBILITY:
Inclusion Criteria:

* Admitted to the BCCH ED with fever (≥38.5 0C) and one or more of the following:

  * cough,
  * runny nose,
  * sore throat, or
  * congested nose.

Exclusion Criteria:

Excluded from the study will be patients who are:

* immuno-compromised,
* have chronic severe respiratory conditions (cystic fibrosis, bronchopulmonary dysplasia),
* chronic heart conditions or
* who is in severe distress requiring immediate care or resuscitation, or
* have had prior assessment in our ED department for the current illness.

Only one child per family can be enrolled.

Ages: 3 Months to 36 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 275 (Estimated)
Dates: Start 2005-12; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Length of Emergency Department visit (from initial physician contact to discharge from Emergency Department)

SECONDARY OUTCOMES:
Rate of antibiotic prescription in Emergency Department.
Rate of ancillary tests performed in Emergency Department.

CONTACTS AND LOCATIONS:
Overall Officials: Eva Thomas, MD, Principal Investigator — The University of British Columbia
Locations (1):
- Children's and Women's Health Centre of BC, Vancouver, British Columbia, Canada